CLINICAL TRIAL: NCT04305821
Title: Intérêt de la protéine S100β Dans Les Traumatismes Crâniens légers Sous Anti-Thrombotiques
Brief Title: Medico-economic Interest of the Protein S100b in Mild Head Trauma Under Anti-thrombotics
Acronym: ISTCAT
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Collaborators: Roche Diagnostics GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: 35RC19_30046_ISTCAT
Record Dates: First submitted 2020-03-10; First posted 2020-03-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Mild Head Injury; Anticoagulant; Antiplatelet
Keywords: Mild head injury, traumatic brain injury, traumatic intracranial hemorrhage; Anticoagulant, antiplatelet, anticoagulant, antithrombotic; S100β protein; health care cost
MeSH Terms: conditions — Brain Injuries, Traumatic; Intracranial Hemorrhage, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Dosage of S100β protein — Dosage of S100β protein

SUMMARY:
Head trauma is a common injury in emergency department. Investigation to search for complication is guided by the clinical examination and the case history, such as taking anti-thrombotics. Cranial computed tomography (CCT) is the gold standard to investigate, and is mandatory in case of antithrombotic drugs.

Recently, some biomarkers have proven their utility to rule-out mild head trauma without CCT in the general population. Among these biomarkers, S100β protein has been added in guidelines for mild head trauma. Some studies have found similar data in population taking anticoagulant or antiplatelet drugs.

The investigators aim to prove medical utility of S100β protein in population under antithrombotics, by the reduction of CCT use. Then, The investigators hypothesize that the add of S100β protein reduces cost of health care in the management of head injury in that population.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old
* Taking antithrombotic medication (antiplatelet drugs, K vitamin antagonist, direct oral anticoagulants, heparins)
* Mild head trauma with Glasgow coma scale ≥ 13
* Trauma occured ≤ 6 hours
* Agreeing the participation in the study

Exclusion Criteria:

* Head injury occured > 6 hours
* Patient < 18 years old or under juridic protection
* pregnant women
* polytrauma
* Glasgow coma scale ≤ 12
* ancient or actual cerebral ou cutaneous neoplasia

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient taking antithrombotic medication with mild head trauma and trauma occured ≤ 6 hours
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Diagnostic performances are evaluated by AUC | 1 day
  Diagnostic performances of S100β protein in case of mild head trauma for detection of traumatic intracranial lesion in patients under antithrombotic medication compare to cranial computed tomography.
Diagnostic performances are evaluated by sensibility, specificity | 1 day
  Diagnostic performances of S100β protein in case of mild head trauma for detection of traumatic intracranial lesion in patients under antithrombotic medication compare to cranial computed tomography.
Diagnostic performances of S100β protein in case of mild head trauma for detection of traumatic intracranial lesion in patients under antithrombotic medication compare to cranial computed tomography. | 1 day
  Diagnostic performances are evaluated by positive and negative predictive values between the strategy with S100β protein compared to the strategy with systematic cranial computed tomography.

CONTACTS AND LOCATIONS:
Overall Officials: Cédric GANGLOFF, MD, Principal Investigator — Centre Hospitalier Univesitaire de Rennes
Locations (1):
- Centre Hospitalier Universitaire de Rennes, Rennes, France